CLINICAL TRIAL: NCT01926626
Title: Evaluation of Moclobemide, a Reversible MAO-A Inhibitor, as an Adjunct to Nicotine Replacement Therapy in Female Smokers
Acronym: RIMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jed E. Rose (Other)
Collaborators: Philip Morris USA, Inc. (Industry); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Jed E. Rose, Professor, Department of Psychiatry and Behavioral Sciences, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00044174; P50DA027840-01 (NIH)
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Results first posted 2015-07-29 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Nicotine Dependence
Keywords: Nicotine addiction; Smoking Cessation; Quit Smoking; moclobemide; Nicotine Patch
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Tobacco Use Cessation Devices; Nicotine; Moclobemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nicotine Patch+Moclobemide (Experimental): After 1 week of pre-cessation nicotine patch treatment (21 mg/24 h patches), participants will receive moclobemide (400 mg/day in 2 divided doses) for 11 weeks, ending 10 weeks after the target quit date. Nicotine patch treatment will continue at 21 mg/24 h for an additional week prior to the quit date, and then for 6 weeks after the quit date, followed by 14 mg/24 h for 2 weeks and 7 mg/24 h for 2 weeks. All treatment will terminate 10 weeks after the quit date.
  Interventions: Drug: Nicotine Patch; Drug: Moclobemide

INTERVENTIONS:
Drug: Nicotine Patch — Pre-Quit Period: 2 weeks of patch use (21mg/24hr)
  Post Quit Period: 10 weeks of patch use (21mg/24hr for 6 weeks, 14mg/24hr for 2 weeks, and 7mg/24hr for 2 weeks)
  Other Names: Nicoderm
Drug: Moclobemide — Pre-Quit Period: 1 week of moclobemide use (400 mg/day in 2 divided doses)
  Post Quit Period: 10 weeks of moclobemide use (400 mg/day in 2 divided doses)
  Other Names: reversible MAO-A inhibitor

SUMMARY:
The proposed study will assess the efficacy of moclobemide, a selective, reversible MAO-A inhibitor, in facilitating smoking cessation in treatment-seeking female smokers. This rationale is based on several findings from previous work: 1) cigarette smoke contains constituents that inhibit both forms of the enzyme monoamine oxidase (MAO-A and MAO-B); 2) that severity of depression symptoms after smoking abstinence is correlated with the level of MAO-A inhibition previously obtained from smoking; 3) moclobemide, an MAO-A inhibitor was found efficacious in a smoking cessation treatment trial (Berlin et al., 1995); and 4) women show a greater association between smoking and depression than men and women smokers in our previous trials report smoking to alleviate symptoms of depression to a greater extent than men.

ELIGIBILITY:
Inclusion Criteria:

* Have no known serious medical conditions;
* Female;
* Are 18-65 years old;
* Smoke an average of at least 20 cigarettes per day;
* Have smoked at least one cumulative year;
* Have a Fagerstrom Test for Nicotine Dependence score of at least 5;
* Have an expired air carbon monoxide (CO) reading of at least 10ppm;
* Able to read and understand English;
* Express a desire to quit smoking in the next thirty days.

Potential subjects must agree to avoid the following during their participation in this study:

* excessive alcohol consumption;
* use of other antidepressants;
* general anesthesia;
* participation in any other nicotine-related modification strategy outside of this protocol;
* use of tobacco products other than cigarettes, including pipe tobacco, cigars, e-cigarettes, snuff, and chewing tobacco;
* use of experimental (investigational) drugs or devices;
* use of illegal drugs;
* cimetidine;
* Tyramine rich foods;
* use of opiate medications.

Exclusion Criteria:

* Hypertension;
* Hypotension with symptoms;
* Coronary heart disease;
* Lifetime history of heart attack;
* Cardiac rhythm disorder;
* Chest pains;
* Cardiac (heart) disorder;
* Active skin disorder;
* Liver or kidney disorder;
* Gastrointestinal problems or disease other than gastroesophageal reflux or heartburn;
* Active ulcers in the past 30 days;
* Currently Symptomatic lung disorder/disease;
* Brain abnormality;
* Migraine headaches that occur more frequently than once per week;
* Recent, unexplained fainting spells;
* Problems giving blood samples;
* Diabetes (unless controlled by diet and exercise alone);
* Current cancer or treatment for cancer in the past six;
* Other major medical condition;
* Current psychiatric disease;
* Suicidal ideation (within the past 10 years) or lifetime occurrence of attempted suicide;
* Current depression;
* Bulimia or anorexia;
* Use (within the past 45 days) of psychiatric medications including antidepressants and anti-psychotics;
* Use (within the past 30 days) of:

  * Illegal drugs (or if the urine drug screen is positive for tetrahydrocannabinol (THC), Cocaine, Amphetamine, Opiates, Methamphetamines, phencyclidine (PCP), Benzodiazepines, or Barbiturates),
  * Experimental (investigational) drugs;
  * Any medications that are known to affect smoking cessation (e.g. clonidine);
  * Smokeless tobacco (chewing tobacco, snuff), pipes or e-cigarettes;
  * Wellbutrin, bupropion, Zyban, Chantix, nicotine replacement therapy or any other smoking cessation aid.
* Use of opiate medications for pain or sleep (non-opiate medication for pain or sleep will be allowed) within the past 14 days;
* Smokes more than one cigar a month.
* Alcohol abuse;
* Significant adverse reaction to nicotine patches, in the past.
* Known hypersensitivity to moclobemide or other MAO-A inhibitors.
* Current participation or recent participation (in the past 30 days) in another smoking study at our center or another research facility.
* Current participation or recent participation (in the past six months) in another medical research study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-09; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jed E Rose, Ph.D., Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Duke Center for Smoking Cessation, Charlotte, North Carolina
  - Duke Center forSmoking Cessation, Durham, North Carolina
  - Duke Center for Smoking Cessation, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 76 participants who were enrolled, 38 participants attended Study Session 1: 1 participant voluntarily withdrew prior to Study Session 1, 3 participants were lost to contact prior to Study Session 1, and 34 were withdrawn from the study by the PI or medical staff because they did not meet inclusion criteria or met exclusion criteria.
Groups:
- Nicotine Patch+Moclobemide: After 1 week of pre-cessation nicotine patch treatment (21 mg/24 h patches), participants will receive moclobemide (400 mg/day in 2 divided doses) for 11 weeks, ending 10 weeks after the target quit date. Nicotine patch treatment will continue at 21 mg/24 h for an additional week prior to the quit date, and then for 6 weeks after the quit date, followed by 14 mg/24 h for 2 weeks and 7 mg/24 h for 2 weeks. All treatment will terminate 10 weeks after the quit date.
  Nicotine Patch: Pre-Quit Period: 2 weeks of patch use (21mg/24hr)
  Post Quit Period: 10 weeks of patch use (21mg/24hr for 6 weeks, 14mg/24hr for 2 weeks, and 7mg/24hr for 2 weeks)
  Moclobemide: Pre-Quit Period: 1 week of moclobemide use (400 mg/day in 2 divided doses)
  Post Quit Period: 10 weeks of moclobemide use (400 mg/day in 2 divided doses)
Period: Overall Study
Arm/Group | Nicotine Patch+Moclobemide
Started | 38
Received Moclobemide | 37
Completed | 16
Not Completed | 22
Not completed — Withdrawal by Subject | 15
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Arm/Group | Nicotine Patch+Moclobemide
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.53 (9.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Continuous Four-week Abstinence From Smoking
Description: Number of participants who reported continuous four-week abstinence from smoking (weeks 6-10 post target quit date), confirmed by expired air carbon monoxide (CO).
Time Frame: Weeks 6-10 post quit day
Measure: Number; unit: participants
Arm/Group | Nicotine Patch+Moclobemide
Number analyzed (Participants) | 38
participants | 7

2. Secondary Outcome: Point Abstinence From Smoking at Six Months Post Quit
Description: Number of participants who reported 7-day point abstinence from smoking at six months post quit, confirmed by expired air CO.
Time Frame: 7 day point abstinence from smoking at six months post quit
Measure: Number; unit: participants
Arm/Group | Nicotine Patch+Moclobemide
Number analyzed (Participants) | 38
participants | 2

3. Secondary Outcome: Continuous Ten Week Abstinence From Smoking
Description: Number of participants who reported continuous ten-week abstinence from smoking (weeks 1-10 post quit day), confirmed by expired air CO.
Time Frame: 10 weeks post quit day
Measure: Number; unit: participants
Arm/Group | Nicotine Patch+Moclobemide
Number analyzed (Participants) | 38
participants | 4

4. Secondary Outcome: Percentage of Change in Smoking Withdrawal Symptoms
Description: Withdrawal symptoms will be assessed by questionnaire on Quit Day, 1 week post quit, 3 weeks post quit, 6 weeks post quit,10 weeks post quit and 6 months post quit (if applicable) using the Shiffman-Jarvik questionnaire, which consists of 33-items rated from 1 to 7, where 1= not at all, 2= very little, 3= a little, 4= moderately, 5= a lot, 6= quite a lot, and 7= extremely. The 33 items are grouped into 8 subscales: Craving, Negative Affect, Appetite, Arousal, Somatic - Anxiety, Somatic - G.I., Somatic - Respiratory Tract, and Habit Withdrawal. The range of scores for each subscale will be 1-7, with higher scores indicating more of the withdrawal symptom having been experienced.
Time Frame: Quit day and 1 week, 3 weeks, 6 weeks, 10 weeks and 6 months post quit day
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | Nicotine Patch+Moclobemide
Number analyzed (Participants) | 38
percentage of change
  Craving -- % change 1 week from Quit Day | -8.07 (7.928)
  Craving -- % change 3 weeks from Quit Day | -13.18 (4.144)
  Craving -- % change 6 weeks from Quit Day | -14.24 (4.63)
  Craving -- % change 10 weeks from Quit Day | -13.41 (6.912)
  Craving -- % change 6 months from Quit Day | 23.71 (63.690)
  Negative Affect -- % change 1 week from Quit Day | -22.82 (4.057)
  Negative Affect -- % change 3 weeks from Quit Day | -14.26 (4.327)
  Negative Affect -- % change 6 weeks from Quit Day | -21.53 (4.051)
  Negative Affect -- % change 10 weeks from Quit Day | -13.92 (4.968)
  Negative Affect -- % change 6 months from Quit Day | 48.87 (65.334)
  Appetite -- % change 1 week from Quit Day | -11.40 (5.486)
  Appetite -- % change 3 weeks from Quit Day | -4.39 (7.881)
  Appetite -- % change 6 weeks from Quit Day | -17.07 (8.819)
  Appetite -- % change 10 weeks from Quit Day | 0.73 (16.033)
  Appetite -- % change 6 months from Quit Day | 27.24 (74.446)
  Arousal -- % change 1 week from Quit Day | 29.81 (8.824)
  Arousal -- % change 3 weeks from Quit Day | 29.03 (7.004)
  Arousal -- % change 6 weeks from Quit Day | 29.99 (6.915)
  Arousal -- % change 10 weeks from Quit Day | 18.95 (6.715)
  Arousal -- % change 6 months from Quit Day | 190.88 (78.496)
  Anxiety -- % change 1 week from Quit Day | -4.65 (3.803)
  Anxiety -- % change 3 weeks from Quit Day | -5.80 (4.788)
  Anxiety -- % change 6 weeks from Quit Day | -4.48 (5.098)
  Anxiety -- % change 10 weeks from Quit Day | -9.44 (6.375)
  Anxiety -- % change 6 months from Quit Day | -38.79 (19.553)
  Gastrointestinal -- % change 1 week from Quit Day | -5.80 (3.365)
  Gastrointestinal -- % change 3 weeks from Quit Day | -2.03 (6.602)
  Gastrointestinal -- % change 6 weeks from Quit Day | 4.55 (16.189)
  Gastrointestinal - % change 10 weeks from Quit Day | -12.20 (5.100)
  Gastrointestinal - % change 6 months from Quit Day | -33.66 (18.204)
  Respiratory -- % change 1 week from Quit Day | 7.26 (6.978)
  Respiratory -- % change 3 weeks from Quit Day | 2.06 (11.161)
  Respiratory -- % change 6 weeks from Quit Day | -5.16 (8.628)
  Respiratory -- % change 10 weeks from Quit Day | -13.28 (8.696)
  Respiratory -- % change 6 months from Quit Day | -38.79 (19.553)
  Habit -- % change 1 week from Quit Day | -9.26 (7.272)
  Habit -- % change 3 weeks from Quit Day | -11.41 (6.309)
  Habit -- % change 6 weeks from Quit Day | -12.22 (7.705)
  Habit -- % change 10 weeks from Quit Day | 1.49 (14.642)
  Habit -- % change 6 months from Quit Day | -38.79 (19.553)

5. Other Pre Specified Outcome: Safety of Moclobemide + Nicotine Patch
Description: Safety of the moclobemide + nicotine patch treatment will be assessed by tabulating the number of participants rating side effects > "moderate".
Time Frame: 1, 2, 4, 7 and 11 weeks after starting Moclobemide + Nicotine Patch
Population: Participants who received Moclobemide.
Measure: Number; unit: participants
Arm/Group | Nicotine Patch+Moclobemide
Number analyzed (Participants) | 37
participants | 21

6. Secondary Outcome: Percentage of Change in Expired Air Carbon Monoxide (CO) During the First Week of Nicotine Patch Treatment.
Description: The initial response to nicotine patch will be assessed by looking at the percent change in expired air carbon monoxide (CO) at the end of week one (Study Visit 2) relative to baseline (Study Visit 1).
Time Frame: Baseline and 1 week
Population: Participants who received Moclobemide.
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | Nicotine Patch+Moclobemide
Number analyzed (Participants) | 37
percentage of change | -18.38 (5.551)

7. Other Pre Specified Outcome: Tolerability of Moclobemide + Nicotine Patch
Description: Tolerability of the moclobemide + nicotine patch treatment will be assessed by tabulating the number of participants requiring dose reductions (or discontinuation of medication).
Time Frame: 1, 2, 4, 7 and 11 weeks after starting Moclobemide + Nicotine Patch
Population: Participants who received Moclobemide.
Measure: Number; unit: participants
Arm/Group | Nicotine Patch+Moclobemide
Number analyzed (Participants) | 37
participants | 17

ADVERSE EVENTS:
Time Frame: Subjects were receiving study drugs for twelve weeks. At each study session during this period subjects completed a questionnaire about side effects. Subjects were also told to contact us between study sessions if side effects were bothersome.
Description: One subject discontinued study participation after the first study session; therefore, no side effects data pertaining to study interventions were collected for this subject.
Arm/Group | Nicotine Patch+Moclobemide
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 29/37
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Patch+Moclobemide (N=37)
Insomnia (Nervous system disorders) | 12 (21)
Tiredness (Nervous system disorders) | 12 (14)
Nightmares (Nervous system disorders) | 5 (5)
Vivid dreams (Nervous system disorders) | 13 (27)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 7 (11)
Excessive sweating (Nervous system disorders) | 4 (14)
Increased appetite (General disorders) | 7 (11)
Loss of appetite (General disorders) | 2 (2)
Altered taste (Nervous system disorders) | 6 (8)
Dry mouth (General disorders) | 9 (18)
Thirst (General disorders) | 10 (19)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Chest Pain (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Heartburn (Gastrointestinal disorders) | 3 (4)
Muscle / joint pain (Musculoskeletal and connective tissue disorders) | 5 (7)
Anxiety (Psychiatric disorders) | 5 (6)
Depression (Psychiatric disorders) | 2 (5)
Agitation / restlessness (Nervous system disorders) | 4 (7)
Itching at patch site (Skin and subcutaneous tissue disorders) | 11 (14)
Rash at patch site (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes